CLINICAL TRIAL: NCT06974305
Title: Investigation of Interictal Metabolic and Electrophysiologic Changes in Epilepsy Through Trimodal Neuroimaging
Brief Title: PET/MRI/EEG Imaging Study in Epilepsy
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ciprian Catana, MD, PhD, Professor of Radiology, Massachusetts General Hospital
Other Study IDs: 2022P000929
Record Dates: First submitted 2024-03-12; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
Keywords: Functional PET; FDG-PET; Functional MRI; EEG; Epilepsy; Neuroimaging; Multimodal imaging
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Healthy control subjects with no major medical history
  Interventions: Radiation: FDG-PET/fMRI/EEG imaging
- Subjects with Epilepsy: Subjects diagnosed with epilepsy and with abnormal electrical activity recorded on interictal EEG.
  Interventions: Radiation: FDG-PET/fMRI/EEG imaging

INTERVENTIONS:
Radiation: FDG-PET/fMRI/EEG imaging — Subject will undergo simultaneous EEG, fMRI, and FDG-PET imaging. This includes the use of a standard injected radioactive marker used in PET imaging.

SUMMARY:
This study aims to better understand how epilepsy alters brain function through neuroimaging of healthy people and people with epilepsy. The study investigates how changes in brain metabolism (sugar consumption, measured by positron emission tomography [FDG-PET], and blood flow, measured by functional magnetic resonance imaging [fMRI]) relate to abnormal interictal electrical activity associated with epilepsy (measured by electroencephalography [EEG]). The study will also compare how the three imaging modalities localize regions of abnormal function in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older

Additional Inclusion Criteria for Subjects with Epilepsy:

* Diagnosed with epilepsy with abnormal interictal EEG

Exclusion Criteria:

* Contraindications to PET, MRI, or EEG imaging
* History of severe brain disease such as stroke and head trauma
* History of brain surgery
* History of type I or II diabetes mellitus
* Fasting plasma glucose level >200 mg/dL
* Employed under direct supervision of the PI conducting the research

Additional Exclusion Criteria for Healthy Subjects:

* Current use of drugs that modulate brain function
* Current or past history of major medical, neurological, or psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study populations are healthy people and people with epilepsy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Image analysis | Image analysis to be performed after imaging sessions are complete.
  There are no interventions in this study and thus no outcome measures. Primary goal of the study will be achieved with image analysis on the PET/MRI/EEG data.

CONTACTS AND LOCATIONS:
Overall Officials: Ciprian Catana, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Athinoula A. Martinos Center, Charlestown, Massachusetts, United States